CLINICAL TRIAL: NCT05976048
Title: Implementation of Actinic Keratosis Guideline Among General Practitioners. Retrospective Cohort Study on Prescription Patterns in the Treatment of Actinic Keratosis.
Brief Title: Implementation of Actinic Keratosis Guideline Among General Practitioners.
Status: Active, not recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-1313
Record Dates: First submitted 2023-07-20; First posted 2023-08-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Actinic Keratoses
Keywords: actinic keratosis; general physician; 5-fluorouracil cream; general practitioner
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study investigates 5-fluorouracil cream prescription trends by general practitioners for the treatment of field changes of actinic keratosis over the years 2016-2021. The aim is to analyse whether the publication of the multidisciplinary guideline on suspect skin lesions for general practitioners in 2017 has made an impact in the prescribing behaviour of general practitioners.

DETAILED DESCRIPTION:
Actinic keratosis is the most common epithelial precancerous lesion among the Caucasian race. With an increase in prevalence worldwide due to an aging population and rise of ultraviolet exposure actinic keratosis are among the most frequently encountered skin lesions in clinical practice. Both dermatologists and general practitioners are increasingly confronted with actinic keratosis, entailing to higher healthcare costs and time burden.

There are many therapeutic modalities for the treatment of actinic keratosis, depending on multiple factors such as distribution, characteristics, patient preference, side effects, availability and costs. Treatment options can be divided into: lesion directed therapy en field directed therapy. Both dermatologists and general practitioners can treat actinic keratosis and 5-fluorouracil cream can also be prescribed by general practitioners.

The objective of this study was to investigate 5-fluorouracil cream prescription trends by general practitioner for the treatment of field changes of actinic keratosis over the years 2016-2021.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* diagnosis actinic keratosis (clinical diagnosed or by biopsy)

Exclusion Criteria:

* cutaneous malignancy (suspicion)
* immunosuppressive co-medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data of patients with actinic keratosis in the general practitioners extracted from the Research network family medicine (RNFM) Maastricht database between 2016 - 2021.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percentage (%) of longitudinal changes in prescriptions of 5-fluorouracil cream | Measurement years 2016, 2019 and 2021
  Percentage (%) of longitudinal changes in prescriptions of 5-fluorouracil cream by general practitioners for the diagnosis actinic keratosis, measured from the Research Network Family Medicine Maastricht database between 2016 - 2021. The Research Network Family Medicine is a registration database with information about the affiliated general practices.

CONTACTS AND LOCATIONS:
Overall Officials: Klara Mosterd, prof.dr., Principal Investigator — Maastricht UMC
Locations (1):
- Ellen Oyen, Maastricht, Netherlands